CLINICAL TRIAL: NCT02731274
Title: Physical Activity and Motor Memory in Pedal Dexterity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Castelo Branco (Other)
Responsible Party: Principal Investigator, André Ramalho, Mss, Instituto Politécnico de Castelo Branco
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESE IPCB02
Record Dates: First submitted 2016-03-23; First posted 2016-04-07 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motor memory consolidation (Experimental): Subjects were divided in two groups: a control group and an experimental one. Before the intervention of physical exercise program, subjects performed a Tapping Pedal Test to measure baseline performance. After the intervention, the assessment of the impact of exercise on motor memory consolidation was held in three stages: Training; 1 hour after training and 24 hours after training.
  Interventions: Other: Regular physical activity in Motor memory consolidation
- Control (No Intervention)

INTERVENTIONS:
Other: Regular physical activity in Motor memory consolidation — After the intervention, the assessment of the impact of exercise on motor memory consolidation was held in three stages: Training; 1 hour after training and 24 hours after training. For the analysis of the results, descriptive and inferential statistics were used.
  Arms: Motor memory consolidation

SUMMARY:
The main purpose of this study was to investigate if a six months period of physical exercise, could improve motor memory consolidation in elderly people on pedal dexterity

DETAILED DESCRIPTION:
34 subjects of both genders, with a mean age of 71 years old participated in the study. Subjects were divided in two groups: a control group and an experimental one. Before the intervention of physical exercise program, subjects performed a Tapping Pedal Test to measure baseline performance. After the intervention, the assessment of the impact of exercise on motor memory consolidation was held in three stages: Training; 1 hour after training and 24 hours after training.

ELIGIBILITY:
Inclusion Criteria:

* individuals not engaged in physical activity;
* persons aged from 65 years.

Exclusion Criteria:

* sensory abnormalities;
* mental abnormalities;
* motor abnormalities;
* other atypical health problems.

Ages: 65 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Subjects performed a Tapping Pedal Test to measure a performance in motor memory consolidation. | 6 months
  investigate if a six months period of physical exercise could improve motor memory consolidation in elderly people

IPD SHARING:
Plan to Share IPD: No